CLINICAL TRIAL: NCT01735786
Title: EndoClotTM Absorbable Polysaccharide Hemostat for Preventing Rbleeding After Endoscopic Mucosal Resection (EMR)
Brief Title: EndoClot for Preventing Rebleeding After Endoscopic Mucosal Resection (EMR)
Status: Completed | Type: Observational
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Zhiguo Liu, Associated Professor, Xijing Hospital of Digestive Diseases
Other Study IDs: 20121125
Record Dates: First submitted 2012-11-25; First posted 2012-11-28 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: Endoscopic Hemostasis; Colonic Polyps
Keywords: Endoscopic Hemostasis; EndoClot Absorbable Polysaccharide Hemostat; Colonic Polyps
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Treatment group: Subjects in this group will received Endoclot treatment immediately after EMR.
  Interventions: Device: EndoClot
- Control group: Subjects in this group will not received any hemostasis treatment after EMR.

INTERVENTIONS:
Device: EndoClot — EndoClot hemostat is applied immediately after EMR to achieve hemostasis.
  Groups: Treatment group

SUMMARY:
Endoscopic mucosal resection (EMR) has been widely used as a diagnostic and treatment techniques of gastrointestinal small lesions. Postoperative rebleeding is one of the common complication following EMR. Several endoscopic hemostasis methods are currently in use. EndoClot® absorbable polysaccharide hemostat (PAPH) as a new hemostasis material was previously used for surgical hemostasis, but the therapeutic effect and safety in endoscopic application remains unknown. This study has been designed to observe the effect of rebleeding prevention after EMR.

ELIGIBILITY:
Inclusion Criteria:

* consecutive cases of colorectal polyps and submucosal lesions with anticipated complete removal endoscopically by EMR.

Exclusion Criteria:

* severe cardiovascular diseases, liver and kidney dysfunction;
* platelet and coagulation dysfunction (PLT < 50*109/L, INR > 2);
* cases that have taken anticoagulant drugs or non-steroidal anti-inflammatory drugs within 1 month before the procedure;
* cases unavailable for follow-up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive cases of colorectal mucosal and submucosal lesions with intented EMR treatment
Sampling Method: Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2010-04; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Rebleeding rate after EMR procedure | up to 1 week
  Rebleeding rate up to 1 week was obtained by clinical manifestations such as melana; decreased hemoglobin > 20g/L; hemodynamic instability or active bleeding from mucosal defect under endoscope.

SECONDARY OUTCOMES:
Mucosal healing after EMR | up to 1 month
  Colonoscopy will be repeated 1 month after EMR procedure to observe if application of Endoclot will delay the musosal healing.
gastrointestinal tract obstruction | up to 1 month
  Gastrointestinal tract obstruction has been previously reported as a possible adverse effect of hemostats, therefore it was observed in the current study.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiguo Liu, M.D., Principal Investigator — Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi, China 710032
Locations (1):
- Xijing Hospital of Digestive Diseases, Xi’an, Shanxi, China